CLINICAL TRIAL: NCT06816199
Title: A Prospective Cohort Study Exploring the Safety and the Efficiency of Hyperbaric Oxygen in Treating Traumatic Brain Injury During Nonacute Phrase
Brief Title: The Safety and the Efficiency of Hyperbaric Oxygen in Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1224
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; hyperbaric oxygen
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-hyperbaric oxygen exposure group: Participants with traumatic brain injuries will always be excluded from hyperbaric oxygen therapy
  Interventions: Other: Hyperbaric oxygen exposure

INTERVENTIONS:
Other: Hyperbaric oxygen exposure — Between 1 week and 3 months after the traumatic brain injury, participants will receive hyperbaric oxygen therapy on a 2.0 ATA protocol for 60 minutes once a day, five times a week.

SUMMARY:
The goal of this observational study is to learn about the safety and long-term effects of hyperbaric oxygen therapy in participants over the age of 18 with traumatic brain injury (TBI).

The main question it aims to answer are:

Does hyperbaric oxygen therapy raise independence in daily living and the ability to engage in social activities in participants with TBI when treated with hyperbaric oxygen therapy during the non-acute phrase after injury? What medical problems do participants have when treated with hyperbaric oxygen therapy? Whether or not participants have used hyperbaric oxygen therapy as part of their routine medical treatment for TBI, they will answer online or telephone survey questions about their functional independence for 2 years.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the safety and long-term effects of hyperbaric oxygen therapy in participants over the age of 18 with traumatic brain injury (TBI). This is a multicenter prospective cohort study.

The main question it aims to answer are:

Does hyperbaric oxygen therapy raise independence in daily living and the ability to engage in social activities in participants with TBI when treated with hyperbaric oxygen therapy during the non-acute phrase after injury? What medical problems do participants have when treated with hyperbaric oxygen therapy? Whether or not participants have used hyperbaric oxygen therapy as part of their routine medical treatment for TBI during non-acute phrase after injury, they will answer online or telephone survey questions about their functional independence (including cognitive functioning, physical disability, mental status, employment and social activities) for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~90 years old
2. Patients with traumatic brain injury admitted to the rehabilitation department meet one of the following indicators:

1) Clear history of exogenous trauma-causing disease (such as car accidents, heavy objects, falls, violent assaults, explosive injuries, etc.) 2) GCS score of 3 to 15 points (excluding all kinds of poisoning, sedation, shock factors) 3. Clear presence of at least one of the following imaging signs on cranial CT or MRI: Traumatic intracranial hemorrhage, subdural hematoma, epidural hematoma, cerebral contusion, ventricular hemorrhage, subarachnoid hemorrhage, or brainstem injury; 4. good compliance, signed informed consent, and those who were judged by the investigator to be eligible for enrollment.

Exclusion Criteria:

1. Sequelae of previous spinal cord injury or combination of spinal cord injury in this injury;
2. Severe coagulation disorders;
3. Pregnancy status;
4. Any other factors that the investigator considers to be a potential risk to the subject or that interfere with the subject.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this observational cohort study, all patients with craniocerebral injuries who satisfy the enrollment requirements and do not meet the exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Extended Glasgow Outcome Scale,GOSE | 6-month, 12-month and 24-month after injury
  Overall functional outcomes for participants with traumatic brain injury

SECONDARY OUTCOMES:
Function Independent Measure, FIM | 6-month, 12-month and 24-month after injury
  This scale is for non-comatose patients after traumatic brain injury and includes motor and cognitive function ratings

OTHER OUTCOMES:
Rivermead Post Concussion Symptoms Questionnaire，RPQ | 6-month, 12-month and 24-month after injury
  Mainly for mild traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Zhang, Principal Investigator — Departments of Physical Medithe Second Affiliated Hospital of Zhejiang University School of Medicine; Sujuan Li, Study Director — Fu Xing Hospital, Capital Medical University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Maas AIR, Menon DK, Manley GT, Abrams M, Akerlund C, Andelic N, Aries M, Bashford T, Bell MJ, Bodien YG, Brett BL, Buki A, Chesnut RM, Citerio G, Clark D, Clasby B, Cooper DJ, Czeiter E, Czosnyka M, Dams-O'Connor K, De Keyser V, Diaz-Arrastia R, Ercole A, van Essen TA, Falvey E, Ferguson AR, Figaji A, Fitzgerald M, Foreman B, Gantner D, Gao G, Giacino J, Gravesteijn B, Guiza F, Gupta D, Gurnell M, Haagsma JA, Hammond FM, Hawryluk G, Hutchinson P, van der Jagt M, Jain S, Jain S, Jiang JY, Kent H, Kolias A, Kompanje EJO, Lecky F, Lingsma HF, Maegele M, Majdan M, Markowitz A, McCrea M, Meyfroidt G, Mikolic A, Mondello S, Mukherjee P, Nelson D, Nelson LD, Newcombe V, Okonkwo D, Oresic M, Peul W, Pisica D, Polinder S, Ponsford J, Puybasset L, Raj R, Robba C, Roe C, Rosand J, Schueler P, Sharp DJ, Smielewski P, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Temkin N, Tenovuo O, Theadom A, Thomas I, Espin AT, Turgeon AF, Unterberg A, Van Praag D, van Veen E, Verheyden J, Vyvere TV, Wang KKW, Wiegers EJA, Williams WH, Wilson L, Wisniewski SR, Younsi A, Yue JK, Yuh EL, Zeiler FA, Zeldovich M, Zemek R; InTBIR Participants and Investigators. Traumatic brain injury: progress and challenges in prevention, clinical care, and research. Lancet Neurol. 2022 Nov;21(11):1004-1060. doi: 10.1016/S1474-4422(22)00309-X. Epub 2022 Sep 29. PMID 36183712
- [Background] Kowalski RG, Hammond FM, Weintraub AH, Nakase-Richardson R, Zafonte RD, Whyte J, Giacino JT. Recovery of Consciousness and Functional Outcome in Moderate and Severe Traumatic Brain Injury. JAMA Neurol. 2021 May 1;78(5):548-557. doi: 10.1001/jamaneurol.2021.0084. PMID 33646273
- [Background] McCrea MA, Giacino JT, Barber J, Temkin NR, Nelson LD, Levin HS, Dikmen S, Stein M, Bodien YG, Boase K, Taylor SR, Vassar M, Mukherjee P, Robertson C, Diaz-Arrastia R, Okonkwo DO, Markowitz AJ, Manley GT; TRACK-TBI Investigators; Adeoye O, Badjatia N, Bullock MR, Chesnut R, Corrigan JD, Crawford K, Duhaime AC, Ellenbogen R, Feeser VR, Ferguson AR, Foreman B, Gardner R, Gaudette E, Goldman D, Gonzalez L, Gopinath S, Gullapalli R, Hemphill JC, Hotz G, Jain S, Keene CD, Korley FK, Kramer J, Kreitzer N, Lindsell C, Machamer J, Madden C, Martin A, McAllister T, Merchant R, Ngwenya LB, Noel F, Nolan A, Palacios E, Perl D, Puccio A, Rabinowitz M, Rosand J, Sander A, Satris G, Schnyer D, Seabury S, Sherer M, Toga A, Valadka A, Wang K, Yue JK, Yuh E, Zafonte R. Functional Outcomes Over the First Year After Moderate to Severe Traumatic Brain Injury in the Prospective, Longitudinal TRACK-TBI Study. JAMA Neurol. 2021 Aug 1;78(8):982-992. doi: 10.1001/jamaneurol.2021.2043. PMID 34228047
- [Background] Schimmel S, El Sayed B, Lockard G, Gordon J, Young I, D'Egidio F, Lee JY, Rodriguez T, Borlongan CV. Identifying the Target Traumatic Brain Injury Population for Hyperbaric Oxygen Therapy. Int J Mol Sci. 2023 Sep 27;24(19):14612. doi: 10.3390/ijms241914612. PMID 37834059